CLINICAL TRIAL: NCT05823233
Title: Investigation of the Effect of Eccentric Stretching on Pain, Grip Strength and Functional Level in Patients With Lateral Epicondylitis
Brief Title: Effect of Eccentric Stretching in Patients With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-161
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Cold application+Deep friction+Home exercise+Eccentric stretching
  Interventions: Other: Cold application+Deep friction+Home exercise+Eccentric stretching
- Control Group (Experimental): Cold application +Deep friction +Home exercise
  Interventions: Other: Cold application+Deep friction+Home exercise

INTERVENTIONS:
Other: Cold application+Deep friction+Home exercise+Eccentric stretching — In our study, deep friction massage will be performed by the researcher with the tip of the thumb, maintaining the pressure for 3-5 minutes in the posterior direction to the tenoosseous junction. The application will be performed 3 times a week for a total of 12 sessions for 4 weeks. After the deep friction massage, cold application will be made for 15 minutes. Simultaneously with the electrical stimulation of the affected arm, the patient will be asked to stretch for 5 seconds and rest for 5 seconds, and doing this 15 times will be considered 1 set. After 1 minute of rest, he will be asked to do this practice for 2 more sets, so 3 sets of 15 repetitions will be completed in total. A total of 12 sessions will be applied 3 days a week for 4 weeks. In our study, a home exercise program consisting of passive stretching and strengthening (concentric and eccentric) exercises will be applied.
  Arms: Study group
Other: Cold application+Deep friction+Home exercise — In our study, deep friction massage will be performed by the researcher with the tip of the thumb, maintaining the pressure for 3-5 minutes in the posterior direction to the tenoosseous junction. The application will be performed 3 times a week for a total of 12 sessions for 4 weeks. After the deep friction massage, cold application will be made for 15 minutes. In our study, a home exercise program consisting of passive stretching and strengthening (concentric and eccentric) exercises will be applied.
  Arms: Control Group

SUMMARY:
Lateral Epicondylitis; is a disease characterized by insidious onset pain in the lateral elbow of the forearm, which radiates to the distal part of the forearm and increases with grip and wrist extension. Pain originates from the origin of the wrist and finger extensors and is more felt during repetitive, forceful wrist extension or pronation and supination, during exercise or occupational use. It is a musculoskeletal lesion. Although it is so common, no consensus has yet been reached regarding its clinic, pathophysiology, and treatment. It is known that the primary etiological factor in the pathology of lateral epicondylitis is the overloading of the aponeurosis of the joint extensor muscles attachment site. Repetitive overuse causes tendon damage with macroscopic abnormalities of tendon collagen. The final stage of tendinopathy is characterized by abnormal tendon structure and degenerative features, including neovascularization. Primary pathological changes occur at the proximal musculotendinous insertion of the Extensor carpi radialis brevis. The currently accepted theory is that the process begins with overuse injuries that lead to small tears of the extensor carpi radialis brevis, sometimes the extensor digitorum communis muscle.

The prevalence of lateral epicondylitis peaks between the ages of 35 and 55, and lateral epicondylitis primarily affects the dominant side. There is no clear consensus on the involvement of men and women, and it appears independent of gender and ethnicity [6-8]. Due to the symptoms experienced, the people's daily life activities are affected and cause loss of workforce.

Conservative therapy is usually the first line of treatment for lateral epicondylitis. Conservative treatment typically includes rest, non-steroidal anti-inflammatory drugs, and physiotherapy and rehabilitation. Physiotherapy and rehabilitation applications include activity modification, orthosis use, cold-hot application, deep friction massage, stretching and strengthening exercises, electrical stimulation, ultrasound, laser, extracorporeal shock wave therapy, and manual therapy. In addition to FTR approaches, invasive procedures such as corticosteroid/botulinum toxin/glucosamine/autologous injections, prolotherapy, acupuncture, and topical nitric oxide application can be used. In cases where conservative treatment is insufficient, surgical applications are used. Although there are many different treatment methods known in the literature, the superiority of a particular approach for the treatment of lateral epicondylitis has not yet been proven and a consensus has not been reached.

It has been known for a long time that eccentric exercises based on the extension of the muscle length can cause damage to the muscle fibers due to stretching and late-onset muscle pain. However, when they are applied in a regular and controlled manner, they adaptively strengthen and protect the muscle tissue. In clinical and animal studies, it has been found that reaching muscle length at an angle greater than the optimum angle of the muscle causes eccentric exercise, which in turn reduces muscle damage and increases joint range of motion.

Although studies continue to understand the mechanisms of post-exercise muscle damage and the protective muscle response that develops after exercise, no study has been found in the literature on eccentric stretching applied to patients with lateral epicondylitis. Therefore, the aim of our study is to investigate the effect of eccentric stretching on pain, grip strength, and functional level in patients with lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 - 65
* Having been diagnosed with Lateral Epicondylitis,
* Pain localized in the elbow for more than 3 months

Exclusion Criteria:

* Those who have had major surgery or trauma related to the musculoskeletal system, especially the elbow region
* Steroid injection to the elbow area in the last 3 months,
* Those with neurological disease
* Those who received physiotherapeutic intervention in the elbow area in the last 3 months
* Having infection and local dermatological problems in the treatment area Those with rheumatic disease in the active period
* Those with systemic diseases (Diabetes, hypothyroidism, infection, malignancy...)
* Those with serious psychological problems (BDI score of 30 and above)
* Pregnancy
* Presence of malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 weeks
  It will be used to objectively determine the degree of pain at rest and during activity. Visual Analogue Scale is a 10 cm line drawn in the horizontal plane on a white sheet of paper. The words "no pain" are on the left end and "the most severe pain you have ever encountered in your life" are on the right. It was explained to the patient that the severity of pain increased from left to right, and he was asked to mark the severity of his own pain separately on this line at rest and during movement. There will be 2 different evaluations as Visual Analogue Scale-Rest and Visual Analogue Scale-Activity. Evaluations will be measured at the start of treatment and at the end of the study.
Grip Strength | 4 weeks
  Grip strength will be measured with the Jamar hand dynamometer while the patient is sitting in a chair with the shoulder in adduction and neutral position, elbow flexed to 90 degrees, forearm and wrist in neutral position. 3 measurements will be made for each patient and 30 seconds of rest will be given between measurements. Patients will be asked for the maximum grip they can achieve and the best result of 3 repetitions will be recorded. Measurement will also be made on the unaffected side and the power difference will be recorded.
Pinchmeter | 4 weeks
  Palmar measurement is evaluated by squeezing the pinch meter with the medial of the thumb and supporting the other fingers from the lateral.
Muscle Tone and Stiffness | 4 weeks
  Muscle tone and stiffness will be evaluated with a myotonometer. The myotonometer was developed for the objective measurement of mechanical muscle properties. Myotonometry reflects the viscoelastic properties of the muscle such as tone and stiffness by creating oscillation in the muscle fiber and is an acceptable and reliable method for measuring the mechanical properties of the muscle. Myotonometer can measure the firmness of tissues 2 cm below the epidermis. MyotonPRO is a new technology for assessing musculoskeletal stiffness; It is widely used in scientific fields.
Patient-Rated Tennis Elbow Evaluation | 4 weeks
  Overend et al. were created to evaluate treatment specifically for lateral epicondylitis patients. Later, it was reorganized by the same study group and named the patient-based tennis elbow evaluation questionnaire (Patient-Rated Tennis Elbow Evaluation). The questionnaire consists of 15 questions questioning the difficulties and pain experienced by the patients with the elbow in the past week. In the first part, the level of pain (5 questions), and in the second part, functions related to the elbow (6 questions about special activities, 4 questions about daily activities) are evaluated. The total score ranges from 0-100, with high scores indicating increased pain and loss of functionality. A high score indicates worsening health. In 2010, Altan et al. The Turkish version was created by Patient-Rated Tennis Elbow Evaluation and it was found to be valid and reliable. The Turkish version of the questionnaire will be used in our study.
Quick Disability of the Arm, Shoulder and Hand Questionnaire | 4 weeks
  Quick Disability of the Arm, Shoulder, and Hand Questionnaire is a short version that can be used to assess disability caused by musculoskeletal problems involving the upper extremity, activity limitation, as well as limitation of leisure time activities and participation in work. In all questions, the patient marks the appropriate answer on the 5-point Likert system (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not doing at all). According to the results of the Disability of the Arm, Shoulder, and Hand Questionnaire and Quick-Disability of the Arm, Shoulder, and Hand Questionnaire; A result between 0-100 is obtained from each section (0 = no excuse, 100 = maximum apology). A high score indicates worsening health.
Nottingham Health Profile:- | 4 weeks
  The Nottingham Health Profile will be used in our quality of life assessment. In the questionnaire consisting of 38 items, 6 different parameters related to health status are evaluated. These parameters are physical activity (8 items), emotional reactions (9 items), energy (3 items), social isolation (5 items), pain (8 items), and sleep (5 items). Each sub-parameter is scored between 0-100. A high score indicates worsening health. The total score is obtained by summing all sub-parameter scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Zeyinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No